CLINICAL TRIAL: NCT05267600
Title: A Phase 2/3, Randomized, Double-Blinded, Placebo-Controlled, Parallel-Group Study to Investigate the Efficacy and Safety of Efgartigimod PH20 SC in Adult Participants With Bullous Pemphigoid
Brief Title: A Phase 2/3 Study of Efgartigimod PH20 SC in Adult Participants With Bullous Pemphigoid
Acronym: BALLAD
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: argenx (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ARGX-113-2009
Record Dates: First submitted 2022-02-14; First posted 2022-03-04 (Actual); Results first posted 2025-10-23 (Actual); Last update posted 2025-10-23 (Actual); Status verified 2025-09

CONDITIONS: Bullous Pemphigoid
MeSH Terms: conditions — Pemphigoid, Bullous | interventions — Prednisone

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- efgartigimod PH20 SC (Experimental): participants receiving efgartigimod PH20 SC on top of Prednisone
  Interventions: Biological: efgartigimod PH20 SC; Drug: Prednisone
- placebo PH20 SC (Placebo Comparator): participants receiving placebo PH20 SC on top of Prednisone
  Interventions: Other: placebo; Drug: Prednisone

INTERVENTIONS:
Biological: efgartigimod PH20 SC — Subcutaneous injection of efgartigimod coformulated with rHuPH20, a permeation enhancer
  Arms: efgartigimod PH20 SC
Other: placebo — Subcutaneous injection of placebo coformulated with rHuPH20, a permeation enhancer
  Arms: placebo PH20 SC
Drug: Prednisone — Oral Prednisone

SUMMARY:
ARGX-113-2009 is an operationally seamless 2-part, phase 2/3, prospective, global, multicenter, randomized, double-blinded, placebo-controlled study to investigate the efficacy, safety, tolerability, immunogenicity, participant-reported outcome measures (including those assessing participant QoL), PK, and PD of efgartigimod PH20 SC administered via subcutaneous (SC) injection in adult participants with moderate to severe BP. This study intends to demonstrate that efgartigimod is an effective and safe treatment for BP, providing participants with control of disease activity (CDA) and eventually remission while reducing their cumulative exposure to OCS.

study will consist of 2 parts:

* Part A of the study is a phase 2 evaluation that intends to provide proof of concept for the therapeutic activity of efgartigimod PH20 SC in participants with BP.
* Part B of the study is a phase 3 evaluation that intends to confirm the results obtained from part A in a separate, larger group of participants with BP.

An interim analysis will be performed during part A (on data obtained through week 26 for all Part A participants) to assess the primary endpoint and several secondary endpoints, confirm the appropriate sample size for part B of the study, and determine whether the efficacy results observed through week 26 of part A warrant continued study of efgartigimod PH20 SC for the treatment of participants with BP (futility analysis).

ELIGIBILITY:
Inclusion Criteria:

* The participant is willing and able to do the following:

  1. understand the requirements of the study
  2. provide written informed consent
  3. comply with the study protocol procedures.
* The participant is male or female and has reached the age of consent at the time of signing the informed consent form (ICF).
* Participants have clinical signs of BP.
* Contraceptive use should be consistent with local regulations regarding the methods of contraception for those participating in clinical studies and: Women of childbearing potential must have a negative serum pregnancy test at screening and a negative urine pregnancy test at baseline before study intervention can be administered.

The full list of inclusion criteria can be found in the protocol.

Exclusion Criteria:

* Other forms of pemphigoid or other autoimmune bullous diseases (AIBDs).
* Received unstable dose of treatments known to cause or exacerbate BP for at least 4 weeks prior to the baseline visit
* Use of BP treatments other than oral corticosteroids (OCS), topical corticosteroids (TCS), conventional immunosuppressants or dapsone.
* Known contraindication to OCS therapy
* Active, chronic or latent infection at screening
* Positive COVID-19 test result at screening (testing performed if required per local regulations).
* History of malignancy unless deemed cured by adequate treatment with no evidence of recurrence for ≥3 years before the first administration of the IMP. Participants with the following cancers can be included at any time, provided they are adequately treated prior to their participation in the study: Basal cell or squamous cell skin cancer, Carcinoma in situ of the cervix, Carcinoma in situ of the breast, Incidental histological finding of prostate cancer
* Clinical evidence of other significant serious diseases, have had a recent surgery, or who have any other condition that, in the opinion of the investigator, could confound the results of the study or put the patient at undue risk or prevent participants from complying with protocol requirements
* Use of an investigational product within 3 months before the first dose of IMP
* Previously participated in a clinical study with efgartigimod or currently participating in another interventional clinical study
* Known hypersensitivity to any of the components of the administered treatments
* Positive serum test at screening for an active infection: HBV, HCV, HIV
* Current or history (ie, within 12 months of screening) of alcohol, drug, or medication abuse as assessed by the investigator
* Pregnant or lactating females and those who intend to become pregnant during the study
* Live or live-attenuated vaccine received <4 weeks before baseline visit

The full list of exclusion criteria can be found in the protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 98 (Actual)
Dates: Start 2022-06-09 (Actual); Primary Completion 2024-09-13 (Actual); Study Completion 2024-09-13 (Actual)

CONTACTS AND LOCATIONS:
Locations (129):
- United States (21):
  - Investigator site 74 - US0010178, Phoenix, Arizona
  - Investigator site 6 - US0010138, Fountain Valley, California
  - Investigator site 121 - US0010092, Redwood City, California
  - Investigator site 72 - US0010186, Santa Monica, California
  - Investigator site 10 - US0010153, Castle Rock, Colorado
  - Investigator site 2 - US0010087, Boca Raton, Florida
  - Investigator site 21 - US0010152, Clearwater, Florida
  - Investigator site 1 - US0010017, Miami, Florida
  - Investigator site 13 - US0010155, West Lafayette, Indiana
  - Investigator site 35 - US0010156, Louisville, Kentucky
  - Investigator site 50 - US0010149, Ann Arbor, Michigan
  - Investigator site 115 - US0010157, Jackson, Mississippi
  - Investigator site 73 - US0010098, St Louis, Missouri
  - Investigator site 85 - US0010159, Lebanon, New Hampshire
  - Investigator site 5 - US0010088, Buffalo, New York
  - Investigator site 93 - US0010169, New York, New York
  - Investigator site 4 - US0010137, Fairborn, Ohio
  - Investigator site 25 - US0010158, Pittsburgh, Pennsylvania
  - Investigator site 34 - US0010182, Houston, Texas
  - Investigator site 92 - US0010150, Murray, Utah
  - Investigator site 3 - US0010151, Morgantown, West Virginia
- Australia (3):
  - Investigator site 36 - AU0610013, Fitzroy
  - Investigator site 27 - AU0610006, Kogarah
  - Investigator site 125 - AU0610019, Woolloongabba
- Bulgaria (3):
  - Investigator site 28 - BG3590018, Sofia
  - Investigator site 14 - BG3590010, Sofia
  - Investigator site 15 - BG3590020, Stara Zagora
- China (15):
  - Investigator site 111 - CN0860064, Beijing
  - Investigator site 91 - CN0860017, Beijing
  - Investigator site 95 - CN0860018, Chengdu
  - Investigator site 116 - CN0860027, Chongqing
  - Investigator site 108 - CN0860023, Fujian
  - Investigator site 107 - CN0860021, Guangzhou
  - Investigator site 110 - CN0860053, Guanzhou
  - Investigator site 128 - CN0860097, Hefei
  - Investigator site 124 - CN0860098, Nanchang
  - Investigator site 94 - CN0860066, Nanyang
  - Investigator site 127 - CN860020, Shanghai
  - Investigator site 123 - CN0860095, Shanghai
  - Investigator site 122 - CN0860065, Ürümqi
  - Investigator site 109 - CN0860025, Wuhan
  - Investigator site 126 - CN0860026, Zhengzhou
- Croatia (3):
  - Investigator site 22 - HR3850003, Split
  - Investigator site 16 - HR3850002, Zagreb
  - Investigator site 37 - HR3850001, Zagreb
- Czechia (4):
  - Investigator site 97 - CZ4200015, Brno
  - Investigator site 118 - CZ4200016, Hradec Králové
  - Investigator site 117 - CZ4200013, Plzen-Bory
  - Investigator site 96 - CZ4200012, Prague
- France (2):
  - Investigator site 38 - FR0330040, Nice
  - Investigator site 29 - FR0330029, Rouen
- Germany (11):
  - Investigator site 46 - DE0490039, Berlin
  - Investigator site 54 - DE0490030, Dresden
  - Investigator site 80 - DE0490041, Düsseldorf
  - Investigator site 57 - DE0490046, Erlangen
  - Investigator site 51 - DE0490008, Essen
  - Investigator site 52 - DE0490024, Frankfurt am Main
  - Investigator site 53 - DE0490023, Freiburg im Breisgau
  - Investigator site 56 - DE0490028, Kiel
  - Investigator site 45 - DE0490001, Marburg
  - Investigator site 75 - DE0490047, München
  - Investigator site 55 - DE0490026, Würzburg
- Greece (6):
  - Investigator site 60 - GE0300004, Athens
  - Investigator site 62 - GE0300006, Athens
  - Investigator site 58 - GR0300001, Athens
  - Investigator site 76 - GR030003, Chaïdári
  - Investigator site 61 - GE0300002, Thessaloniki
  - Investigator site 59 - GR0300005, Thessaloniki
- Hungary (3):
  - Investigator site 26 - HU0360023, Budapest
  - Investigator site 11 - HU0360003, Debrecen
  - Investigator site 7 - HU0360008, Pécs
- Israel (4):
  - Investigator site 39 - IL9720003, Afula
  - Investigator site 63 - IL9720018, Haifa
  - Investigator site 41 - IL9720001, Ramat Gan
  - Investigator site 40 - IL9720002, Tel Aviv
- Italy (12):
  - Investigator site 65 - IT0390055, Bologna
  - Investigator site 43 - IT0390060, Brescia
  - Investigator site 78 - IT0390039, Catania
  - Investigator site 47 - IT0390031, Florence
  - Investigator site 86 - IT0390067, Florence
  - Investigator site 81 - IT0390030, Genova
  - Investigator site 77 - IT0390062, Milan
  - Investigator site 119 - IT0390066, Parma
  - Investigator site 64 - IT0390061, Pavia
  - Investigator site 23 - IT0390006, Roma
  - Investigator site 42 - IT0390005, Roma
  - Investigator site 30 - IT0390040, Siena
- Japan (11):
  - Investigator site 103 - JP0810070, Kumamoto
  - Investigator site 99 - JP0810050, Kurume
  - Investigator site 104 - JP0810071, Maebashi
  - Investigator site 100 - JP0810046, Nagakute
  - Investigator site 129 - JP0810073, Niigata
  - Investigator site 101 - JP0810049, Osaka
  - Investigator site 102 - JP0810069, Ōsaka-sayama
  - Investigator site 112 - JP0810045, Sapporo
  - Investigator site 105 - JP0810067, Sendai
  - Investigator site 98 - JP0810043, Tokyo
  - Investigator site 106 - JP0810068, Yokohama
- Latvia (3):
  - Investigator site 87 - LV3710005, Riga
  - Investigator site 82 - LV3710003, Riga
  - Investigator site 88 - LV3710004, Riga
- Investigator site 66 - NL0310015, Groningen, Netherlands
- Poland (5):
  - Investigator site 17 - PL0480047, Lodz
  - Investigator site 79 - PL0480025, Rzeszów
  - Investigator site 83 - PL0480050, Warsaw
  - Investigator site 18 - PL0480048, Wroclaw
  - Investigator site 19 - PL0480046, Wroclaw
- Romania (2):
  - Investigator site 90 - RO0400014, Cluj-Napoca
  - Investigator site 89 - RO0400015, Iași
- Serbia (4):
  - Investigator 68 - RS381011, Belgrade
  - Investigator site 84 - RS3810010, Belgrade
  - Investigator site 67 - RS3810012, Niš
  - Investigator site 69 - RS3810009, Novi Sad
- Slovakia (3):
  - Investigator site 113 - SK4210002, Bratislava
  - Investigator site 120 - SK4210004, Košice
  - Investigator site 114 - SK4210003, Trnava
- Spain (10):
  - Investigator site 32 - ES0340050, Badalona
  - Investigator 24 - ES0340051, Barcelona
  - Investigator site 8 - ES0340053, Granada
  - Investigator site 12 - ES0340025, Madrid
  - Investigator 20 - ES0340029, Madrid
  - Investigator site 49 - ES0340058, Manises
  - Investigator site 31 - ES0340057, Málaga
  - Investigator site 48 - ES0340059, Mieres
  - Investigator site 9 - ES0340052, Seville
  - Investigator site 70 - ES0340061, Valencia
- United Kingdom (3):
  - Investigator site 33 - UK0440022, Bristol
  - Investigator site 71 - UK0440036, London
  - Investigator site 44 - UK0440037, Southampton

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Parts A and B were identical in schedule, structure, eligibility requirements, assessments, and conduct therefore the results are shown with the pooled data from part A and part B.
Groups:
- Efgartigimod PH20 SC: All participants from Part A and Part B receiving efgartigimod PH20 SC. Participants received concurrent oral prednisone (or equivalent) at a starting dose of 0.5 mg/kg/day. The dose of prednisone was adjusted according to recommendations as per protocol.
- Placebo PH20 SC: All participants from Part A and Part B receiving placebo PH20 SC. Participants received concurrent oral prednisone (or equivalent) at a starting dose of 0.5 mg/kg/day. The dose of prednisone was adjusted according to recommendations as per protocol.
Period: Overall Study
Arm/Group | Efgartigimod PH20 SC | Placebo PH20 SC
Started | 50 | 48
Completed | 35 | 35
Not Completed | 15 | 13
Not completed — Adverse Event | 1 | 4
Not completed — Death | 1 | 2
Not completed — Lack of Efficacy | 1 | 2
Not completed — Lost to Follow-up | 3 | 0
Not completed — Physician Decision | 4 | 0
Not completed — Treatment Unblinded | 0 | 1
Not completed — Withdrawal by Subject | 5 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Efgartigimod PH20 SC | Placebo PH20 SC | Total
Number analyzed (Participants) | 50 | 48 | 98
Age, Continuous [Mean (Standard Deviation); unit: years] | 71.0 (12.02) | 70.9 (9.37) | 70.9 (10.75)
Age, Customized [Count of Participants; unit: Participants]
  18 - <65 years | 12 | 11 | 23
  65 - <75 years | 18 | 17 | 35
  75 - <85 years | 15 | 17 | 32
  >=85 years | 5 | 3 | 8
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 37 | 35 | 72
  Male | 13 | 13 | 26
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  AMERICAN INDIAN OR ALASKA NATIVE | 1 | 0 | 1
  ASIAN | 8 | 9 | 17
  MULTIPLE | 1 | 0 | 1
  WHITE | 40 | 39 | 79
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  HISPANIC OR LATINO | 1 | 0 | 1
  NOT HISPANIC OR LATINO | 49 | 48 | 97

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With CRoff at Week 36
Description: CRoff = complete remission while receiving efgartigimod PH20 SC or placebo and being off oral corticosteroid therapy for at least 8 weeks. Complete remission is defined as the absence of new lesions, complete healing of existing lesions and absence of pruritus.
Time Frame: at week 36
Measure: Count of Participants; unit: Participants
Arm/Group | Efgartigimod PH20 SC | Placebo PH20 SC
Number analyzed (Participants) | 50 | 48
Participants | 8 | 2

2. Secondary Outcome: Cumulative OCS Dose
Description: OCS = oral corticosteroid
Time Frame: up to week 36
Measure: Mean (Standard Deviation); unit: mg/kg/day
Arm/Group | Efgartigimod PH20 SC | Placebo PH20 SC
Number analyzed (Participants) | 50 | 48
mg/kg/day | 0.242 (0.138) | 0.289 (0.173)

3. Secondary Outcome: Number of Participants Who Achieve an IGA-BP Score of 0 While Off OCS Therapy for ≥8 Weeks at Week 36
Description: IGA-BP = Investigator Global Assessment of Bullous Pemphigoid. IGA-BP scores range from 0-4, with a higher score representing severe BP. OCS = oral corticosteroid
Time Frame: at week 36
Measure: Count of Participants; unit: Participants
Arm/Group | Efgartigimod PH20 SC | Placebo PH20 SC
Number analyzed (Participants) | 50 | 48
Participants | 9 | 3

4. Secondary Outcome: Number of Participants With CDA Who Remained Free of Relapse Through Week 36
Description: Control of disease activity (CDA) is defined as the point at which new lesions ceased to form, established lesions began to heal, and pruritic symptoms started to abate. Relapse is defined as the appearance of 3 or more new lesions a month or at least 1 large lesion that did not heal within 1 week, or extension of established lesions or daily pruritus in a participant who had achieved CDA.
Time Frame: up to week 36
Measure: Count of Participants; unit: Participants
Arm/Group | Efgartigimod PH20 SC | Placebo PH20 SC
Number analyzed (Participants) | 50 | 48
Participants | 7 | 8

5. Secondary Outcome: Number of Participants With CRmin at Week 36
Description: CRmin = complete remission receiving minimal oral corticosteroids for at least 8 weeks. Minimal oral corticosteroid (OCS) therapy is defined as ≤0.1 mg/kg/day of prednisone (or equivalent).
Time Frame: at week 36
Measure: Count of Participants; unit: Participants
Arm/Group | Efgartigimod PH20 SC | Placebo PH20 SC
Number analyzed (Participants) | 50 | 48
Participants | 8 | 3

6. Secondary Outcome: Change From Baseline to Week 36 in the 24-Hour Average Itch NRS Score
Description: Itch NRS = Itch Numerical Rating Scale. The Itch NRS scores range from 0-10 with 10 representing the worst imaginable itch.
Time Frame: up to week 36
Population: Only participants with an assessment at baseline and at week 36 are reported.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Efgartigimod PH20 SC | Placebo PH20 SC
Number analyzed (Participants) | 19 | 19
score on a scale | -4.4 (3.35) | -2.4 (4.26)

7. Secondary Outcome: Changes From Baseline in the BPDAI Total Activity Score
Description: BPDAI = Bullous Pemphigoid Disease Area Index (BPDAI) Total Activity Score is a tool to objectively measure disease activity. BPDAI scores range from 0 to 360 with a higher score indicating more severe disease (max 240 for total skin activity and 120 for mucosal activity).
Time Frame: up to week 36
Population: Only participants with an assessment at baseline and week 36 are reported here.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Efgartigimod PH20 SC | Placebo PH20 SC
Number analyzed (Participants) | 22 | 19
score on a scale | -43.13 (19.633) | -43.56 (32.584)

8. Secondary Outcome: Time to CDA
Description: CDA = control of disease activity, the point at which new lesions ceased to form, established lesions began to heal, and pruritic symptoms started to abate.
Time Frame: up to week 36
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Efgartigimod PH20 SC | Placebo PH20 SC
Number analyzed (Participants) | 48 | 47
days | 16.0 [10.0 to 17.0] | 15.0 [13.0 to 22.0]

9. Secondary Outcome: Time to CR
Description: CR = complete remission, the absence of new lesions, complete healing of existing lesions, and absence of pruritus.
Time Frame: up to week 36
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Efgartigimod PH20 SC | Placebo PH20 SC
Number analyzed (Participants) | 50 | 48
days | 134.0 [85.0 to NA] — The 95% CI could not be reported because of insufficient number of participants with events | 99.0 [57.0 to 225.0]

10. Secondary Outcome: Time to CRmin
Description: CRmin = complete remission, the absence of new lesions, complete healing of existing lesions, and absence of pruritus while being on minimal dose of OCS for ≥8 Weeks. OCS = oral corticosteroid. Minimal OCS therapy is defined as an oral prednisone dosage of ≤0.10 mg/kg/day (or equivalent).
Time Frame: up to week 36
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Efgartigimod PH20 SC | Placebo PH20 SC
Number analyzed (Participants) | 50 | 48
days | NA [247.0 to NA] — The median and 95% CI could not be reported because of insufficient number of participants with event | NA [NA to NA] — The median and 95% CI could not be reported because of insufficient number of participants with event

11. Secondary Outcome: Time to CRoff/PRoff
Description: CRoff= complete remission (the absence of new lesions, complete healing of existing lesions, and absence of pruritus) while receiving efgartigimod PH20 SC or placebo and being off oral corticosteroid therapy for at least 8 weeks. PRoff = partial remission (the presence of only new transient lesions) while receiving efgartigimod PH20 SC or placebo and being off oral corticosteroid therapy for at least 8 weeks.
Time Frame: up to week 36
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Efgartigimod PH20 SC | Placebo PH20 SC
Number analyzed (Participants) | 50 | 48
days | NA [NA to NA] — The median and 95% CI could not be reported because of insufficient number of participants with events | NA [NA to NA] — The median and 95% CI could not be reported because of insufficient number of participants with events

12. Secondary Outcome: Time to CRoff
Description: CRoff is defined as the absence of new lesions, complete healing of existing lesions, and absence of pruritus while being off OCS therapy for ≥8 weeks.
Time Frame: up to week 36
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Efgartigimod PH20 SC | Placebo PH20 SC
Number analyzed (Participants) | 50 | 48
days | NA [NA to NA] — The median and 95% CI could not be reported because of insufficient number of participants with events | NA [NA to NA] — The median and 95% CI could not be reported because of insufficient number of participants with events

13. Secondary Outcome: Time From CDA to Achieve Relapse
Description: CDA is defined as the point at which new lesions ceased to form, established lesions began to heal, and pruritic symptoms started to abate. Relapse is defined as the appearance of 3 or more new lesions a month or at least 1 large lesion that did not heal within 1 week, or extension of established lesions or daily pruritus in a participant who had achieved CDA.
Time Frame: up to week 36
Population: Only participants achieving CDA are included in this section.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Efgartigimod PH20 SC | Placebo PH20 SC
Number analyzed (Participants) | 48 | 42
days | 114.0 [78.0 to 160.0] | 105.0 [71.0 to 163.0]

14. Secondary Outcome: Number of Participants Who Receive Rescue Therapy Before Week 36
Time Frame: at week 36
Measure: Count of Participants; unit: Participants
Arm/Group | Efgartigimod PH20 SC | Placebo PH20 SC
Number analyzed (Participants) | 50 | 48
Participants | 19 | 18

15. Secondary Outcome: The AIS From the GTI
Description: The Aggregate Improvement Score (AIS) from the Glucocorticoid Toxicity Index (GTI) can range from -346 to 439 with a higher score representing greater corticosteroid toxicity. If a study drug is effective at lowering greater corticosteroid toxicity over time, the score will be lower.
Time Frame: up to week 36
Population: Only participants with a GTI assessment at baseline and at week 36 are reported here.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Efgartigimod PH20 SC | Placebo PH20 SC
Number analyzed (Participants) | 21 | 19
score on a scale | 5.7 (56.98) | 10.9 (45.42)

16. Secondary Outcome: The CWS From the GTI
Description: The Cumulative Worsening Score (CWS) from the Glucocorticoid Toxicity Index (GTI) can range from 0 to 439 with a higher score representing greater corticosteroid toxicity.
Time Frame: up to week 36
Population: Only participants with a GTI assessment at baseline and at week 36 are reported here.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Efgartigimod PH20 SC | Placebo PH20 SC
Number analyzed (Participants) | 21 | 19
score on a scale | 56.1 (40.71) | 47.5 (46.68)

17. Secondary Outcome: EQ-5D-5L VAS Scores Over Time
Description: The EuroQol 5-Dimension 5-Level Visual Analog Scale (EQ-5D-5L VAS) scores range from 0-100 with 0 representing the worst health.
Time Frame: up to week 36
Population: Only participants with an assessment at baseline and at week 36 are reported here.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Efgartigimod PH20 SC | Placebo PH20 SC
Number analyzed (Participants) | 19 | 19
score on a scale | 12.7 (15.94) | 4.5 (24.44)

18. Secondary Outcome: DLQI Scores Over Time
Description: Dermatology Life Quality Index (DLQI) assess the participant's perception of the impact of skin diseases on different aspects of their health-related QoL. Scores range from 0 to 30 with a higher score representing a worse quality of life.
Time Frame: up to week 36
Population: Only participants with an assessment at baseline and at week 36 are reported here.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Efgartigimod PH20 SC | Placebo PH20 SC
Number analyzed (Participants) | 19 | 19
score on a scale | -7.3 (6.25) | -6.7 (7.14)

19. Secondary Outcome: ABQoL Scores Over Time
Description: Autoimmune Bullous Disease Quality of Life Index (ABQoL) questionnaire assesses the impact of Autoimmune Bullous Disease and their therapies on the daily life of patients. Scores range from 0 to 51 with a higher score representing a worse quality of life.
Time Frame: up to week 36
Population: Only participants with an assessment at baseline and at week 36 are analyzed.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Efgartigimod PH20 SC | Placebo PH20 SC
Number analyzed (Participants) | 19 | 19
score on a scale | -12.3 (6.44) | -12.0 (10.92)

20. Secondary Outcome: Efgartigimod Serum Concentrations
Time Frame: up to week 36
Population: The number analyzed differs from overall number analyzed because the following samples were excluded from analysis: Pre-dose samples that were taken after dosing on that day, samples taken outside the visit window, and when the study drug administration prior to the sample is missed.
Measure: Mean (Standard Deviation); unit: ug/mL
Arm/Group | Efgartigimod PH20 SC
Number analyzed (Participants) | 50
ug/mL
  Week 1: number analyzed (Participants) | 46
  Week 1 | 35.7 (13.6)
  Day 10: number analyzed (Participants) | 10
  Day 10 | 96.4 (23.9)
  Week 2: number analyzed (Participants) | 46
  Week 2 | 37.3 (12.5)
  Week 4: number analyzed (Participants) | 42
  Week 4 | 26.0 (11.0)
  Week 8: number analyzed (Participants) | 41
  Week 8 | 25.8 (10.5)
  Week 12: number analyzed (Participants) | 39
  Week 12 | 24.4 (8.92)
  Week 16: number analyzed (Participants) | 35
  Week 16 | 24.3 (8.51)
  Week 20: number analyzed (Participants) | 34
  Week 20 | 23.9 (9.12)
  Week 24: number analyzed (Participants) | 32
  Week 24 | 24.3 (9.98)
  Week 26: number analyzed (Participants) | 27
  Week 26 | 24.6 (10.2)
  Week 28: number analyzed (Participants) | 25
  Week 28 | 23.3 (10.3)
  Week 32: number analyzed (Participants) | 25
  Week 32 | 26.1 (11.3)
  Week 36: number analyzed (Participants) | 17
  Week 36 | 22.2 (8.59)

21. Secondary Outcome: Percent Change of Total IgG Serum Levels From Baseline Over Time
Time Frame: up to 36 weeks
Population: Only participants with an assessment at baseline and at week 36 are reported here.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Efgartigimod PH20 SC | Placebo PH20 SC
Number analyzed (Participants) | 36 | 34
percent change | -46.91 (42.244) | -7.65 (25.374)

22. Secondary Outcome: Percent Change of Anti-BP180 and Anti-BP230 Antibodies From Baseline Over Time
Time Frame: up to 36 weeks
Population: Only participants with an assessment at baseline and at week 36 are reported here (31+34 with values for anti-BP180 and 11+12 with values for anti-BP230).
Measure: Mean (Standard Deviation); unit: Percent change in RU/mL
Arm/Group | Efgartigimod PH20 SC | Placebo PH20 SC
Number analyzed (Participants) | 31 | 34
Percent change in RU/mL
  Percent change of Anti-BP180 antibodies from baseline over time | -58.58 (56.983) | -57.98 (33.470)
  Percent change of Anti-BP230 antibodies from baseline over time: number analyzed (Participants) | 11 | 12
  Percent change of Anti-BP230 antibodies from baseline over time | -46.72 (35.950) | -50.95 (28.617)

23. Secondary Outcome: Incidence of Antidrug Antibodies Against Efgartigimod and Antibodies Produced Against rHuPH20
Time Frame: up to 46 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Efgartigimod PH20 SC | Placebo PH20 SC
Number analyzed (Participants) | 50 | 48
Participants
  ADA against efgartigimod | 2 | 2
  Antibodies against rHuPH20 | 9 | 0

24. Secondary Outcome: Number of Participants (or Their Caregivers) Who Are Determined by Site Staff to be Sufficiently Competent in (Self-)Administering Efgartigimod PH20 SC
Time Frame: up to week 32
Population: The number analyzed for participants and caregivers is the total number who received training and therefore were eligible to be assessed for this outcome (5+4 participants received training and 2+3 caregivers received training).
Measure: Count of Participants; unit: Participants
Arm/Group | Efgartigimod PH20 SC | Placebo PH20 SC
Number analyzed (Participants) | 8 | 18
Participants
  Participants | 5 | 4
  Caregivers: number analyzed (Participants) | 5 | 4
  Caregivers | 2 | 3

ADVERSE EVENTS:
Time Frame: up to 46 weeks
Description: Adverse events were assessed during participant visits.
Arm/Group | Efgartigimod PH20 SC | Placebo PH20 SC
All-Cause Mortality (participants affected / at risk) | 1/50 | 2/48
Serious Adverse Events (participants affected / at risk) | 12/50 | 12/48
Other Adverse Events (participants affected / at risk) | 47/50 | 46/48
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Efgartigimod PH20 SC (N=50) | Placebo PH20 SC (N=48)
ANAEMIA (Blood and lymphatic system disorders) | 1 | 0
ACUTE MYOCARDIAL INFARCTION (Cardiac disorders) | 0 | 1
ATRIAL FIBRILLATION (Cardiac disorders) | 1 | 1
CARDIAC ARREST (Cardiac disorders) | 1 | 0
CARDIAC FAILURE (Cardiac disorders) | 0 | 1
CARDIAC FAILURE ACUTE (Cardiac disorders) | 1 | 0
CARDIAC FAILURE CONGESTIVE (Cardiac disorders) | 1 | 0
COR PULMONALE (Cardiac disorders) | 1 | 0
CORONARY ARTERY STENOSIS (Cardiac disorders) | 0 | 1
SINUS NODE DYSFUNCTION (Cardiac disorders) | 0 | 1
CUSHING'S SYNDROME (Endocrine disorders) | 0 | 1
LENS DISLOCATION (Eye disorders) | 1 | 0
INGUINAL HERNIA (Gastrointestinal disorders) | 1 | 0
INTESTINAL MASS (Gastrointestinal disorders) | 1 | 0
ASTHENIA (General disorders) | 1 | 0
CONDITION AGGRAVATED (General disorders) | 2 | 0
NON-CARDIAC CHEST PAIN (General disorders) | 0 | 1
CELLULITIS GANGRENOUS (Infections and infestations) | 0 | 1
PNEUMONIA (Infections and infestations) | 2 | 0
PNEUMONIA ASPIRATION (Infections and infestations) | 0 | 1
SEPTIC SHOCK (Infections and infestations) | 0 | 1
ANKLE FRACTURE (Injury, poisoning and procedural complications) | 1 | 0
FALL (Injury, poisoning and procedural complications) | 0 | 1
FEMUR FRACTURE (Injury, poisoning and procedural complications) | 1 | 0
MULTIPLE INJURIES (Injury, poisoning and procedural complications) | 0 | 1
SKIN LACERATION (Injury, poisoning and procedural complications) | 1 | 0
STRESS FRACTURE (Injury, poisoning and procedural complications) | 1 | 0
THORACIC VERTEBRAL FRACTURE (Injury, poisoning and procedural complications) | 1 | 0
VASCULAR GRAFT OCCLUSION (Injury, poisoning and procedural complications) | 1 | 0
DEHYDRATION (Metabolism and nutrition disorders) | 0 | 1
DIABETIC KETOACIDOSIS (Metabolism and nutrition disorders) | 0 | 1
OVARIAN EPITHELIAL CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
CAROTID ARTERY OCCLUSION (Nervous system disorders) | 1 | 0
CEREBROVASCULAR DISORDER (Nervous system disorders) | 0 | 1
ENCEPHALOPATHY (Nervous system disorders) | 1 | 0
HYPOTONIA (Nervous system disorders) | 0 | 1
ISCHAEMIC STROKE (Nervous system disorders) | 1 | 0
ACUTE RESPIRATORY FAILURE (Respiratory, thoracic and mediastinal disorders) | 1 | 0
CHRONIC OBSTRUCTIVE PULMONARY DISEASE (Respiratory, thoracic and mediastinal disorders) | 1 | 0
PULMONARY EMBOLISM (Respiratory, thoracic and mediastinal disorders) | 0 | 1
RESPIRATORY FAILURE (Respiratory, thoracic and mediastinal disorders) | 1 | 0
SKIN ULCER (Skin and subcutaneous tissue disorders) | 1 | 0
DEEP VEIN THROMBOSIS (Vascular disorders) | 0 | 2
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Efgartigimod PH20 SC (N=50) | Placebo PH20 SC (N=48)
INCREASED TENDENCY TO BRUISE (Blood and lymphatic system disorders) | 5 | 7
LEUKOCYTOSIS (Blood and lymphatic system disorders) | 0 | 4
LYMPHOPENIA (Blood and lymphatic system disorders) | 5 | 3
CUSHINGOID (Endocrine disorders) | 4 | 0
CONSTIPATION (Gastrointestinal disorders) | 3 | 0
DIARRHOEA (Gastrointestinal disorders) | 5 | 3
NAUSEA (Gastrointestinal disorders) | 3 | 1
VOMITING (Gastrointestinal disorders) | 2 | 4
CONDITION AGGRAVATED (General disorders) | 3 | 0
FATIGUE (General disorders) | 4 | 1
INJECTION SITE ERYTHEMA (General disorders) | 4 | 2
INJECTION SITE PARAESTHESIA (General disorders) | 3 | 2
OEDEMA (General disorders) | 3 | 0
OEDEMA PERIPHERAL (General disorders) | 5 | 5
COVID-19 (Infections and infestations) | 2 | 4
NASOPHARYNGITIS (Infections and infestations) | 3 | 1
PNEUMONIA (Infections and infestations) | 3 | 0
URINARY TRACT INFECTION (Infections and infestations) | 5 | 6
FALL (Injury, poisoning and procedural complications) | 2 | 4
ALANINE AMINOTRANSFERASE INCREASED (Investigations) | 1 | 3
GLYCOSYLATED HAEMOGLOBIN INCREASED (Investigations) | 4 | 3
DIABETES MELLITUS (Metabolism and nutrition disorders) | 3 | 2
HYPOKALAEMIA (Metabolism and nutrition disorders) | 0 | 3
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 4 | 3
BACK PAIN (Musculoskeletal and connective tissue disorders) | 5 | 5
MUSCLE SPASMS (Musculoskeletal and connective tissue disorders) | 3 | 1
MUSCULAR WEAKNESS (Musculoskeletal and connective tissue disorders) | 3 | 0
MYOPATHY (Musculoskeletal and connective tissue disorders) | 3 | 4
DIZZINESS (Nervous system disorders) | 4 | 2
HEADACHE (Nervous system disorders) | 7 | 2
DEPRESSION (Psychiatric disorders) | 5 | 1
INSOMNIA (Psychiatric disorders) | 7 | 8
MANIA (Psychiatric disorders) | 1 | 3
CHRONIC KIDNEY DISEASE (Renal and urinary disorders) | 0 | 3
GLYCOSURIA (Renal and urinary disorders) | 0 | 3
COUGH (Respiratory, thoracic and mediastinal disorders) | 6 | 0
DRY SKIN (Skin and subcutaneous tissue disorders) | 2 | 3
HIRSUTISM (Skin and subcutaneous tissue disorders) | 1 | 3
INTERTRIGO (Skin and subcutaneous tissue disorders) | 4 | 0
PRURITUS (Skin and subcutaneous tissue disorders) | 4 | 5
HYPERTENSION (Vascular disorders) | 6 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2024-02-27): https://cdn.clinicaltrials.gov/large-docs/00/NCT05267600/Prot_000.pdf
  • Statistical Analysis Plan (2024-11-04): https://cdn.clinicaltrials.gov/large-docs/00/NCT05267600/SAP_001.pdf